CLINICAL TRIAL: NCT04346420
Title: Impact of the Double-Trunk Mask on Oxygenation Titration in Patients With COVID-19
Brief Title: Impact of the Double-Trunk Mask on Oxygenation Titration in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Poncin, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DTM-001
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID; Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O2 DTM+ (Experimental): The standard nasal cannula interface is accompanied with the DTM
  Interventions: Device: Double-Trunk Mask
- O2 DTM- (Active Comparator): The standard interface for administering oxygen (nasal cannula or oxygen mask) is worn by the patient, without the DTM
  Interventions: Other: Standard interface

INTERVENTIONS:
Other: Standard interface — The standard interface for administering oxygen (nasal cannula or oxygen mask) is worn by the patient. Oxygen output is adapted to reach a SpO2 target of 94%.
  Arms: O2 DTM-
Device: Double-Trunk Mask — The standard nasal cannula interface accompanied with the DTM is worn by the patient. Oxygen output is adapted to reach a SpO2 target of 94%.
  Arms: O2 DTM+

SUMMARY:
This study will investigate the impact of the Double-Trunk Mask (DTM) on the reduction of oxygen titration in patients with severe hypoxemia.

DETAILED DESCRIPTION:
The Double-Trunk Mask (DTM) is a device designed to increase the fraction of inspired oxygen in patients who receive oxygen therapy. The mask is composed of a regular aerosol mask with corrugated tubing (15 cm length) inserted into two lateral holes.

Each included patient will wear standard nasal cannula in addition to the Double-Trunk Mask for 30 minutes, then only their standard oxygen interface for the next 30 minutes. While maintaining the oxygen saturation by pulse oximetry (SpO2) at a target value of 94%, the impact of the DTM will be assessed by measuring the change of oxygen flow given to the patient.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19
* SpO2 between 92 and 96% with low-flow oxygen therapy (< 15 L/min).

Exclusion Criteria:

* Chronic obstructive pulmonary disease or other chronic respiratory disease
* Confusion
* Hypoxemia corrected (SpO2 ≥ 96%) with O2 flow ≤ 3 L/min
* Contra-indications to arterial blood gas sampling (peripheral arteriopathy, bleeding disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in O2 output | At baseline and 30 minutes after wearing both systems
  The O2 output will be adjusted to maintain a SpO2 of 94% using both systems for administering O2. The O2 flow will be read from the position of the ball in flow meters.

SECONDARY OUTCOMES:
Comfort with the interfaces | 30 minutes after wearing both systems
  A Likert scale from 0 to 5 will be used to measure the subjective comfort of the patient while wearing the standard interface for administering O2 and/or the DTM
Changes in PaO2 | At baseline and 30 minutes after wearing DTM
  Oxygen tension (PaO2) in mmHg will be analyzed from a sample taken from the arterial system
Changes in PaCO2 | At baseline and 30 minutes after wearing DTM
  Carbon dioxide tension (PaCO2) in mmHg will be analyzed from a sample taken from the arterial system.
Changes in pH | At baseline and 30 minutes after wearing DTM
  Potential of Hydrogen (pH) will be analyzed from a sample taken from the arterial system.
Changes in respiratory rate | At baseline and 30 minutes after wearing both systems
  Respiratory rate is measured during one minute by visual inspection.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium